CLINICAL TRIAL: NCT02688465
Title: Effect of an Apomorphine Pump on the Quality of Sleep in Parkinson's Disease Patients (POMPRENELLE).
Acronym: POMPRENELLE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHH_2016_01
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apomorphine pump (Experimental)
  Interventions: Drug: Apomorphine

INTERVENTIONS:
Drug: Apomorphine

SUMMARY:
Parkinson's disease is not only a pathology of movements. There are many non-motor symptoms that complicate and impair patients' quality of life. Among those disorders are sleep disorders.

Insomnia is the most frequent symptom. Most patients report 2-5 awakenings per night and long periods of awakening which occupy 30 to 40% of their night.

Apomorphine is a dopamine agonist that may be administered with a pump . The objective of the study is to assess changes in the quality of sleep in Parkinson's disease patients treated with an apomorphine pump.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients for whom a treatment with an apomorphine pump is indicated

Exclusion Criteria:

* atypical parkinsonian syndrome
* cognitive impairment
* pregnancy
* breast feeding
* patient under a legal protection procedure
* patient denying to participate to the study
* lack of affiliation to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Difference between the Parkinson's disease sleeping disorders (PDSD-2) score before treatment with an apomorphine pump and 3 months after the beginning of the treatment | Three months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation ophtalmique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No